CLINICAL TRIAL: NCT05684250
Title: Effect of Biofeedback Training on Accommodation During Multifocal Lens Wear in Young Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: State University of New York College of Optometry (Other)
Collaborators: William G. & Helen C. Hoffman Foundation (Unknown)
Responsible Party: Principal Investigator, Xiaoying Zhu, OD, PhD, MD, MS, FAAO, Associate Clinical Professor, State University of New York College of Optometry
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRBNET.ORG 1933308
Record Dates: First submitted 2023-01-01; First posted 2023-01-13 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Accomodation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The time course group (Experimental): The time course of the effect of biofeedback training in young adults wearing MFCLs. Subjects will receive one episode of auditory biofeedback training and accommodation will be measured before the training and after the training on a weekly basis for 3 weeks.
  Interventions: Behavioral: Auditory biofeedback training
- The repetition group (Experimental): Subjects will receive one episode of auditory biofeedback training every week for 3 weeks and accommodation will be measured before the training and after the training on a weekly basis.
  Interventions: Behavioral: Auditory biofeedback training
- The longer duration group (Experimental): Subjects will receive one episode of auditory biofeedback training for twice as long every week for 3 weeks and accommodation will be measured before the training and after the training on a weekly basis.
  Interventions: Behavioral: Auditory biofeedback training

INTERVENTIONS:
Behavioral: Auditory biofeedback training — For the auditory biofeedback training, subjects are provided with two tones while fixating a target, one tone related to their accommodative response and the second to the target distance. Their task is to match these tones.

SUMMARY:
This study will examine the accommodative behavior in young adults wearing multifocal soft contact lenses. undergoing myopia control treatments. Subjects will undergo auditory biofeedback training while wearing the multifocal contact lenses to improve the accommodative. This pilot study is divided into three separate experiments and aims to assess:

1. the time course of the effect of biofeedback training in young adults wearing MFCLs -- the time course group
2. whether repeated biofeedback training increases the efficacy in young adults wearing MFCLs -- the repetition group
3. whether a longer training duration, given repeatedly, increases the efficacy in young adults wearing MFCLs -- the longer duration group

The results of this study will be used to design a larger clinical trial to investigate whether increasing accommodative responses through the multifocal contact lenses increases multifocal lenses' treatment effect on myopia management in children.

DETAILED DESCRIPTION:
The public health systems worldwide might soon face an increase in highly myopic patients and with this a rising number of cases with severe eye diseases. By 2050, about five billion people are expected to be myopic and one billion might suffer from a myopia of more than -5 D. According to the World Health Organization, myopia is one of the top factors leading to avoidable blindness. For decades, researchers have been investigating the etiology of this refractive error as well as methods to prevent its progression in children myopic. Among the currently available treatments to slow myopia progression, optical interventions were shown to be a promising and feasible non-invasive approach. Hyperopic retinal defocus is known to induce ocular axial elongation and may be a factor in the progression of myopia. Positive defocus has been shown to reduce axial elongation and contact lenses with bi- or multifocal power profiles that add positive power to the central distance have been used to reduce myopia progression in children. Clinical trial outcomes show progression to be reduced, on average, by 38% on average, but with variable results. This variability may be related to the ways patients accommodate through the lenses. An earlier study found that children wearing multifocal lenses may under-accommodate at near, which could reduce the efficacy of the lenses.

Biofeedback training has been used to change accommodation. Earlier studies attempted to reduce accommodation based on the hypothesis that functional myopia results from a spasm of the ciliary muscle. In contrast, a recent study with young adult myopes successfully applied auditory biofeedback training to *increase* accommodation accuracy and reduce the accommodative lag in individuals by 0.3 D or more at different dioptric distances and while myopic subjects wore multifocal contact lenses. If accommodation was increased by means of auditory biofeedback training in myopic children wearing multifocal soft contact lenses, the treatment efficacy of the lenses might be improved.

The purpose of this pilot study is to investigate whether the frequency and duration of auditory biofeedback training affect their efficacy in increasing accommodative responses through the multifocal lenses.

• STUDY POPULATION

Thirty subjects will be randomized to one of the three study groups:

1. The time course group: The time course of the effect of biofeedback training (one episode) on accommodation in young adults wearing MFCLs will be measured weekly
2. The repetition group: The effect of repeated biofeedback training (one episode per week for 3 weeks) on accommodation through the MFCLs will be measured weekly
3. The longer duration group: The effect of repeated biofeedback training with longer duration (one episode per week for 3 weeks) on accommodation through the MFCLs will be measured weekly

INCLUSION CRITERIA

* Best corrected monocular Snellen visual acuity (VA) ≧ 20/25
* Age 18 to 30 years
* Refractive error spherical equivalent between -0.75 D and -10 D
* Astigmatism ≤ 0.75 D
* Age-appropriate amplitude of accommodation
* No suspected or confirmed eye disease (anamnesis)
* No accommodative or binocular function abnormalities
* Agreement to participate in the study (informed consent of subjects)

EXCLUSION CRITERIA

* Persons who are incapable of giving consent
* Refractive error spherical equivalent < -10 D and > -0.75 D
* Astigmatism > 0.75 D
* Abnormal binocular functions
* Medication affecting accommodative response or causing dry eye

ELIGIBILITY:
Inclusion Criteria:

* Best corrected monocular Snellen visual acuity (VA) ≧ 20/25
* Age 18 to 30 years
* Refractive error spherical equivalent between -0.75 D and -10 D
* Astigmatism ≤ 0.75 D
* Age-appropriate amplitude of accommodation
* No suspected or confirmed eye disease (anamnesis)
* No accommodative or binocular function abnormalities
* Agreement to participate in the study (informed consent of subjects)

Exclusion Criteria:

* Persons who are incapable of giving consent
* Refractive error spherical equivalent < -10 D and > -0.75 D
* Astigmatism > 0.75 D
* Abnormal binocular functions
* Medication affecting accommodative response or causing dry eye

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-07-19 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Accommodation | Immediately before and after one episode of auditory biofeedback training. Change in accommodation from the baseline will be assessed weekly for 3 weeks.
  Accommodative response to 0, 2.5, 3, and 4 D while subjects wear multifocal contact lenses are measured using an infrared powerrefractor.

CONTACTS AND LOCATIONS:
Locations (1):
- State University of New York, College of Optometry, New York, New York, United States